CLINICAL TRIAL: NCT03468764
Title: Evaluation of Hemodynamic Changes Induced by Alveolar Recruitment Maneuver With Respect to Volemic State in Patients Undergoing Anesthesia for Colon Surgery
Brief Title: Hemodynamic Changes Induced by Alveolar Recruitment Maneuver With Respect to Volemic State in Colon Surgery
Acronym: RecruVol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Gemma, Principal Investigator, IRCCS San Raffaele
Other Study IDs: 1/int/2018
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Hypovolemia
Keywords: anesthesia; hemodynamic management; lung recruitment maneuver; hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vigileo monitoring during lung recruitment maneuver — Standard monitoring parameters, invasive blood pressure and hemodynamic values (SVV and CO, through Vigileo device) will be monitored. With the patient in a supine position and as SVV reaches a value of 12-15%, a LRM is performed, consisting in the application of 30 cm H2O continuous positive airway pressure for 30 seconds.
  The alterations in the above mentioned parameters will be registered before and after the maneuver.
  The same procedure will be performed after a 8 ml/kg crystalloids fluid challenge, as soon as SVV reaches the value of 10%.

SUMMARY:
Intraoperative hemodynamic management is important, since even mild variations in circulatory volume can be extremely damaging for patients.

Minimally invasive hemodynamic monitoring are not always available or cost-effective, therefore management of fluids is challenging for anesthesiologists.

This study aims to assess if, after performance of a lung recruitment maneuver (LRM), standard parameter's variation differs between hypovolemic and normovolemic patients.

Patients' volemic state will be assessed with the Vigileo system. Standard monitoring values (heart rate, invasive blood pressure and saturation) will be registered before and after LRMs.

A fluid challenge will be performed and the above mentioned parameters will be recorded again, after a second LRM.

The study is a prospective observational study.

DETAILED DESCRIPTION:
During general anesthesia, it's important to maintain normovolemia, since hypovolemia can cause inadequate tissue perfusion and hypervolemia increases the rate of complications, overall mortality and morbidity.

Critically ill patients commonly present with important hypotension that, in the majority of cases, is promptly treated with intravenous fluids to reverse organ hypoperfusion.

However, previous studies have demonstrated that only 50% of hemodynamically unstable patients are responsive to fluid administration.

In the last decade, attention has been focused on finding a parameter capable of assessing fluid responsiveness in a hypotensive patient.

Recent articles have demonstrated that standard monitoring parameters have no significance for this purpose, while hemodynamic parameters, like stroke volume variation (SVV) or pulse pressure variation (PVV) may have an important role.

An interesting field of research involves heart-lung interactions during mechanical ventilation. In particular, lung recruitment maneuver (LRM) induce physiological cardiovascular alterations and may have a correlation with the volemic state of the patient.

LRMs are commonly performed and safe procedures that consist in application of a continuous positive pressure in the lungs of mechanically ventilated patient, with the aim of improving pulmonary compliance.

The goal of our study is to verify whether the alterations induced by lung recruitment maneuver on commonly registered intraoperative parameters, such as heart rate and arterial blood pressure, actually differ when the maneuver is applied to hypovolemic and normovolemic patients respectively.

Patients undergoing scheduled laparoscopic colon surgery will be enrolled. Informed consent will be obtained during the preoperative anesthesiological visit.

General anaesthesia will be managed according to standard clinical practice. Invasive blood pressure monitoring will be started with a peripheral arterial catheter and hemodynamic parameters (SVV and CO) will be monitored through the Vigileo device.

During the resection phase, the patient has to be maintained in hypovolemic conditions. When SVV reaches a value of 12-15%, a LRM is performed, consisting in the application of 30 cm H2O continuous positive airway pressure for 30 seconds.

Standard monitoring values (heart rate, invasive blood pressure and saturation) will be registered.

Thereafter, a fluid challenge will be performed, consisting in intravenous administration of 8 ml/kg of saline solution over 20 minutes. As soon as SVV will reach a value of 10%, LRM will be performed again and the abovementioned three sets of measurements will be carried out once again.

As standard management of LRM, the maneuver will be stopped if the heart rate would lower below 35 bpm or the systolic blood pressure would lower below 60 mmHg.

The information provided by the study is of interest in cases in which the deployment of sophisticated monitoring, as the Vigileo system, is not feasible or cost-effective. In this way, hemodynamic management during major surgeries would become faster and easier, relying on traditional monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective surgery
* ASA score 1-2-3
* Informed consent

Exclusion Criteria:

* Pregnancy
* Relevant cardiac/pulmonary comorbidities
* Cardiac/kidney failure
* Haemodynamic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled laparoscopic colon surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Hypovolemic indicator | Intraoperative
  Finding an hypovolemic indicator among standard monitoring parameters

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gemma, MD, Study Chair — IRCCS San Raffaele, Milan, Italy
Locations (1):
- S. Raffaele Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No